CLINICAL TRIAL: NCT05132933
Title: Gas Exchange Derangement Physiopathology and Response to Different Levels of Positive End-expiratory Pressure in Critically Ill Patients With COVID-19
Brief Title: Gas Exchange Derangement Physiopathology in Critically Ill Patients With COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Giacomo Grasselli, MD, Professor, Policlinico Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19-SHUNT
Record Dates: First submitted 2021-11-23; First posted 2021-11-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2021-11

CONDITIONS: Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Shunt-group (Experimental): Test of three different levels of positive end-expiratory pressure (PEEP)
  Interventions: Procedure: PEEP trial - Electrical Impedance Tomography

INTERVENTIONS:
Procedure: PEEP trial - Electrical Impedance Tomography — Three different levels of PEEP and two different levels of FiO2 will be tested without changing anything else in the baseline patient ventilation

SUMMARY:
The study was designed to understand the pathophysiology of gas exchange derangement in critically ill patients with COVID-19. Specifically we will evaluate the effect of 3 different levels of positive end-expiratory pressure (PEEP) and two different levels of inspiratory oxygen fraction (FiO2) on gas exchange by analyzing shunt and dead space. Furthermore, complete respiratory mechanics and distribution of ventilation and perfusion by electrical impedance tomography will be assessed at each level of PEEP.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted in intensive care unit for COVID-19 related Acute Respiratory Distress Syndrome (ARDS) requiring invasive mechanical ventilation

Exclusion Criteria:

* Pregnancy
* Hemodynamic instability (80-90 mmHg increase or 30-40 mmHg decrease systolic arterial pressure compared to baseline value or need of vasopressors to maintain systolic blood pressure higher than 85 mmHg or electrocardiogram evidence of ischemia/arrhythmias)
* Presence of pneumothorax and/or pneumomediastinum
* Contraindications to Electrical Impedance Tomography (pacemaker, implantable cardioverter defibrillator, thoracic drainages)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Shunt at three different levels of positive end expiratory pressure (PEEP) | 30 minutes after change of positive end expiratory pressure (PEEP) level
  Shunt measured by arterial and mixed venous blood samples at each level of PEEP

SECONDARY OUTCOMES:
Dead space at three different levels of positive end expiratory pressure (PEEP) | 30 minutes after change of positive end expiratory pressure (PEEP) level
  Dead space measured by capnography at each level of PEEP
Shunt and dead space at two different levels of inspiratory oxygen fraction for each level of positive end expiratory pressure (PEEP) | 30 minutes after change of positive end expiratory pressure (PEEP) level
  Shunt measured by arterial and mixed venous blood samples and dead space measured by capnography at each level of PEEP
Ventilation/perfusion at three different levels of positive end expiratory pressure (PEEP) assessed by electrical impedance tomography (EIT) | 30 minutes after change of positive end expiratory pressure (PEEP) level
  Ventilation/perfusion assessed by Electrical Impedance Tomography at each level of PEEP
Respiratory mechanics at three different levels of positive end expiratory pressure (PEEP) | 30 minutes after change of positive end expiratory pressure (PEEP) level
  Respiratory mechanics (including esophageal pressure measurement) assessed at each level of PEEP by performing end-inspiratory and end-expiratory pauses

CONTACTS AND LOCATIONS:
Overall Officials: Giacomo Grasselli, Professor, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Ospedale Maggiore Policlinico, Milan, MI, Italy

REFERENCES:
- [Derived] Florio G, Zanella A, Slobod D, Guzzardella A, Protti I, Carlesso E, Canakoglu A, Fumagalli J, Scaravilli V, Colombo SM, Caccioppola A, Brioni M, Pesenti AM, Grasselli G. Impact of Positive End-Expiratory Pressure and FiO2 on Lung Mechanics and Intrapulmonary Shunt in Mechanically Ventilated Patients with ARDS Due to COVID-19 Pneumonia. J Intensive Care Med. 2024 May;39(5):420-428. doi: 10.1177/08850666231210485. Epub 2023 Nov 5. PMID 37926984